CLINICAL TRIAL: NCT03717610
Title: Feasibility of Intraoperative Given Hyperthermic Intraperitoneal Chemotherapy (HIPEC) With Cisplatin During a Cytoreductive Surgery in Patients With Recurrent Ovarian, Peritoneal or Fallopian Tube Cancers
Brief Title: Hyperthermic Intraperitoneal Chemotherapy for Treatment of Relapsed Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Marta Lomnytska, Principal Investigator, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 077/2018
Record Dates: First submitted 2018-10-08; First posted 2018-10-24 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete cytoreductive surgery plus HIPEC with cis-platinum100mg/m2 for 90 min (Experimental)
  Interventions: Procedure: radical surgery with HIPEC

INTERVENTIONS:
Procedure: radical surgery with HIPEC — Straight after macroscopic radical cytoreductive surgery, an intraperitoneal hyperthermic perfusion using the open-abdomen technique will be performed with a single dose of cisplatin 100 mg/m2 administered for 90 minutes in the hyperthermic phase (41°C-43°C).

SUMMARY:
This is a feasibility single-center study to investigate the tolerability, toxicity, quality of life, morbidity, mortality of the HIPEC treatment following cytoreductive surgery for treatment of recurrent ovarian, peritoneal, and fallopian tube cancers.

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of gynecological cancer mortality; it is in 75% of cases detected at advanced stages. The standard treatment is cytoreductive surgery with removal of macroscopic tumor, and intravenous chemotherapy. Three randomized trials observed survival gain for ovarian cancer patients that received intraperitoneal chemotherapy after the optimal cytoreduction, however catheter-related complications made the procedure not feasible. A "one-time" hyperthermic intraperitoneal chemotherapy, HIPEC, is an established for peritoneal carcinosis in colorectal cancer, and recently two phase III randomised clinical studies observe survival gain also for ovarian cancer patients after surgery with HIPEC.

Here the investigators, plan to investigate the HIPEC procedure following cytoreductive surgery for recurrent ovarian cancer, a progressed disease without any standard treatment established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of recurrent epithelial ovarian carcinoma, peritoneal carcinoma, or fallopian tube carcinoma after 6 month since platinum-based chemotherapy (first recurrence) and are scheduled for secondary surgical evaluation/cytoreduction
* ECOG/WHO Performance score of 0 to 1
* Adequate respiratory, hepatic, cardiac, kidney and bone marrow function ( Hb >= 8 g/dl, absolute neutrophil count > 1500/mm3, platelets > 100,000/mm3, creatinine clearance > 60 mL/min according to Cockroft formula)
* Adequate renal function Creatinine ≤ 1.5 mg/dl, and adequate hepatic function Bilirubin ≤ 1.5 mg/dl and AST and ALT ≤ 80 IU/L
* Histological types feature would be serous, endometrioid, clear cell, undifferentiated carcinomas, transitional cell carcinoma, or mixed epithelial carcinoma
* No end organ function
* Patients must have less than or equal to 2.5 mm residual disease at the completion of the cytoreductive surgery to be eligible for the study
* Patient-compliant and psychologically able to follow the trial procedures, signature of informed consent.

Exclusion Criteria:

* Evidence of extensive retroperitoneal lymph node disease
* Neuropsychiatric disorders;
* Pregnancy or breast feeding.
* Subjects who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded
* Subjects with invasive malignancies or had any evidence of the other cancer present within the last 3 years. Prior radiation for localized cancer of the breast, head and neck, or skin are permitted, provided that it was completed more than 3 years prior to enrollment, and the subject remains free of recurrent or metastatic disease
* Subjects with active infection that requires parenteral antibiotics
* Tumors of low malignant potential, or non-invasive borderline tumors
* Patients with any underlying cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions, chronic or latent infectious diseases, immune deficiency, or history, which in the opinion of the investigator, places the patient at an unacceptable risk for participation in the study
* Patient with extra-abdominal metastatic disease
* Known platinum (carboplatin or cisplatin) allergy
* Life expectancy < 3 months
* Still, it will not be considered for the HIPEC protocol those patients with unresectable disease (presence of invasive peritoneal implants inoperable or at high risk for resection in critical locations such as hepatic hilum, the mesenteric root, trunk celiac, mesentery, and several small implants the serosa of the small intestine) and / or with residual disease after cytoreduction greater than or equal to 2.5 mm (CC-2 and CC-3).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related toxicities | 3 months after surgery
  Registration of the effects according to NCI CTCAEv4.0 guidelines.

SECONDARY OUTCOMES:
Assessment of quality of life | before surgery, and 4 weeks, 3 months and 6 months after surgery
  EORTC C30 quality of life questionnaire
Assessment of quality of life in relation to ovarian cancer | before surgery, and 4 weeks, 3 months and 6 months after surgery
  EORTC OV28 quality of life questionnaire
Assessment of quality of Life in relation to eventually performed intestinal surgery | before surgery, and 4 weeks, 3 months and 6 months after surgery
  EORTC CR29 quality of life questionnaire
Morbidity | 30 days after surgery
  Rate of the high-grade 3 and 4 complications, according to the Clawien-Dindo scale
Mortality | 90 days after surgery
  Number of participants with lethal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marta Lomnytska, MD, PhD, Principal Investigator — Uppsala University, Sweden
Locations (1):
- Uppsala University Hopsital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No